CLINICAL TRIAL: NCT05519800
Title: The Metabolic Effects of Ultra-endurance Exercise and Training Under Low or High Glycaemic Index-carbohydrate Diets.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: U1111-1281-5048
Record Dates: First submitted 2022-08-15; First posted 2022-08-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: A Randomised Counter-balanced Intervention Study in Endurance Athletes
MeSH Terms: interventions — isomaltulose; maltodextrin

STUDY DESIGN:
Intervention Model Description: randomised counter-balanced
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Glycaemic Index (Active Comparator): A diet comprising of High Glycaemic Carbohydrate. Supplemented with a maltodextrin containing beverage.
  Interventions: Dietary Supplement: Maltodextrin
- Low Glycaemic Index (Experimental): A diet comprising of Low Glycaemic Carbohydrate. Supplemented with an Isomaltulose containing beverage.
  Interventions: Dietary Supplement: Isomaltulose

INTERVENTIONS:
Dietary Supplement: Isomaltulose — Diet will be supplemented with a beverage containing Isomaltulose as a carbohydrate source.
  Other Names: Palatinose
  Arms: Low Glycaemic Index
Dietary Supplement: Maltodextrin — Diet will be supplemented using a beverage containing Maltodextrin.
  Arms: High Glycaemic Index

SUMMARY:
A randomised counter-balanced intervention study in endurance athletes

DETAILED DESCRIPTION:
To characterise glycaemic, dietary, physiological, and metabolic responses around intense endurance exercise and training in ultra-endurance athletes.

Primary objective

• Detail the proportion of time spent in glycaemic ranges over a prolonged period of training under the influence of different GI diets in Ultra-endurance athletes.

Secondary Objectives

* Characterise physiological responses to differing GI diets during a period of extensive endurance exercise through hormonal markers.
* Observe the influence of differing GI diets on the impact of endurance performance and short term recovery from endurance exercise, detailing the influence of different GI carbohydrate on the restoration of performance output.
* Observe the perception of wellness and gut discomfort using either high or low GI diets supplemented with high or low GI carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Male or female aged 18-65 years (both inclusive)
* Otherwise healthy (as judged by premedical questionnaire) and participating in regular training (volume in training >10 h training per week) and participating in endurance events and/or VO2max > 55 ml.kg-1.min-1.

Exclusion Criteria:

* Receipt of any investigational medicinal product within 1 month prior to screening in this trial
* Haemoglobin <8.0 mmol/L (male) or <7.0 mmol/L (female).
* Systemic (oral or i.v.) corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, growth hormone and non-routine vitamins and herbal products. Furthermore, thyroid hormones are not allowed unless the use of these has been stable during the past 3 months.
* Suffer from or history of a life-threatening disease (i.e. cancer judged not to be in full remission except basal cell skin cancer or squamous cell skin cancer), or clinically severe diseases that directly influence the study results, as judged by the Investigator. This does not prohibit the participation of patients taking medications that influences their metabolism (e.g. statin) or cardio- respiratory system (e.g. asthma spray) as long as the therapy is stable and is not adapted throughout the run of the trial. Furthermore, it does not exclude patients how have coeliac disease (or similar diseases or allergies), as long as the disease is stable, and patients are able to stay on their specific (e.g.) gluten- free diet.
* Known cardiac problems defined as decompensated heart failure (New York Heart Association (NYHA) class III and IV) 10 at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time
* Supine blood pressure at screening (after resting for 5 min in supine position) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic (excluding white-coat hypertension; therefore, if a repeated measurement on a second screening Visit shows values within the range, the participant can be included in the trial). This exclusion criterion also pertains to participants being on anti-hypertensives.
* History of clinically significant abnormal ECG issues, as judged by the Investigator.
* Severe retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
* Any chronic disorder or severe disease which, in the opinion of the Investigator might jeopardise participant's safety or compliance with the protocol.
* History of allergies and/or intolerances to drugs or foods or a history of severe anaphylactic reaction e.g. fructose intolerance.
* Significant history of alcoholism or drug/chemical abuse as per Investigator's judgement or a positive result in the urine drug/alcohol screen at the screening Visit.
* Smoker (defined as a participant who is smoking more than 5 cigarettes or the equivalent per day).
* Not able or willing to refrain from smoking or use of nicotine substitute products during the monitoring period.
* Participant with mental incapacity or language barriers precluding adequate understanding or cooperation or who, in the opinion of their general practitioner or the Investigator, should not participate in the trial.
* Participating in any other research trial which may interfere with the current study.
* Potentially non-compliant or uncooperative during the trial, as judged by the Investigator.
* Any condition that would interfere with trial participation or evaluation of results, as judged by the Investigator.
* Any known history of diabetes mellitus, or the use of any anti- hyperglycaemic drug or insulin to treat diabetes and related conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Interstitial Glucose Percentage Coefficient of Variation. | 24 months
  A metric which is related to the daily variation of Interstitial Glucose concentration relative to mean concentration.

SECONDARY OUTCOMES:
Mean blood and interstitial glucose concentration. | 24 Months
  A measure of mean concentration of glucose in both blood and interstitial fluid.
% Time Spent in Range | 24 Months
  A characterisation of Interstitial Glucose Concentration in defined ranges.Hyperglycaemia (+7 mmol.L-1), Euglycaemia (4.0-7 mmol.L-1), Hypoglycaemia (<3.9 mmol.L-1).
Performance changes | 24 Months
  Physical performance as measured by time to task failure following re-feed protocol of either high or low glycaemic carbohydrates
Cardio vascular indicators during exercise | 24 Months
  Observing potential changes in the following during repeated exercise trial. Heart rate Vo2 Fuel Oxidization Carbohydrate:Fat oxidization
Metabolic and hormonal change in response to re-feed of high or low glycaemic carbohydrate. | 24 Months
  Observing any potential adaptation or impact on metabolic or hormones. Assessed through the following Insulin response Intestinal fatty-acid binding protein (iFABP) Triglycerides Glycerol Free Fatty Acids Liver stress enzymes (Alkaline Phosphatase, Aspartate aminotransferase, Alanine transaminase, Gamma-glutamyl transferase & total bilirubin) Cardiac and Muscle enzymes (Heart-type fatty acid binding protein, Cardiac troponin, Creatine kinase & Myoglobin) Ketones
Gut distress | 24 Months
  Record of potential gut distress via Gastrointestinal Symptom Rating Scale (GSRS).
3. Comparison of lifestyle and wellness when on either high or low Glycaemic diet. | 24 months
  Observing impact or changes on daily background activity and sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea Univeristy, Swansea, United Kingdom